CLINICAL TRIAL: NCT02314845
Title: Optimizing Intraoperative Mechanical Ventilation Using EIT-titrated PEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Joaquim Edson Vieira, Associate Professor, Anesthesiology, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAAE_13768713.0.0000.0068
Record Dates: First submitted 2014-11-07; First posted 2014-12-11 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Pulmonary Atelectasis
Keywords: Pulmonary Atelectasis; Pulmonary Ventilation; Anesthesia, General; Electric Impedance; Tomography, Spiral Computed; Intraoperative Period
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optimal PEEP (Experimental): Patients submitted to general anesthesia and abdominal laparoscopic surgery (number=10) or open surgery (number=10) will be submitted to a recruitment maneuver followed by a PEEP titration procedure using Electrical Impedance Tomography (EIT). Patients will be mechanically ventilated during intraoperative period using "Optimal PEEP" determined by Electrical Impedance and FIO2 of 0.5.
  Interventions: Other: Optimal PEEP
- Low PEEP (Other): Patients submitted to general anesthesia and abdominal laparoscopic surgery (number=10) or open surgery (number=10) will be submitted to a recruitment maneuver followed by a PEEP titration procedure EIT. In this arm, the ventilator will be set with a PEEP=4 cmH2O ("Low PEEP") and FIO2 of 0.5 during intraoperative period.
  Interventions: Other: Low PEEP

INTERVENTIONS:
Other: Optimal PEEP — "Optimal PEEP" determined by EIT during a PEEP titration procedure.
  Arms: Optimal PEEP
Other: Low PEEP — Use of PEEP of 4 cmH2O during intraoperative period
  Arms: Low PEEP

SUMMARY:
The purpose of this randomized single center study is to determine the individual PEEP value that produces the best possible compromise of lung collapse and lung hyperdistention. Patients submitted to general anesthesia and mechanical ventilation during surgery (laparoscopy and open surgery) will participate. A PEEP titration procedure will be performed and the "optimal PEEP" value will be determined by electrical impedance tomography (EIT). An ultrasound will be used to record each step of the PEEP titration procedure in a sub-sample of patients. A total of 40 patients will be mechanically ventilated using physiological tidal volume (TV=6mL/kg of IBW) and fraction of inspired oxygen (FIO2) of 0.5 and will be randomized to one of two groups: "optimal PEEP" or a "low PEEP" (4cmH2O). Lung collapse and mechanics will be monitored by EIT throughout the intraoperative period. After extubation, a lung CT will be performed to evaluate the amount of lung collapse.

DETAILED DESCRIPTION:
Patients submitted to general anesthesia and mechanical ventilation commonly develop pulmonary atelectasis, which can cause adverse consequences either intraoperatively or postoperatively. The use of lower, more physiological tidal volumes (6-8 mL/Kg of ideal body weight) during the intraoperative period can minimize the risk of lung injury but may be associated with increased atelectasis. The application of PEEP can prevent the formation of atelectasis and minimize the resulting complications, but at the present time, there is no consensus on how to tailor the level of PEEP to best suit each patient.

Electrical Impedance Tomography (EIT) is a portable non-invasive monitor that enables the analysis of lung function in a continuous mode.

The aim of this study is to evaluate the use of Electrical Impedance Tomography (EIT), in the intraoperative period, as a tool for selecting "optimal PEEP" using a PEEP titration procedure, as well as assessing the evolution of pulmonary function during this period.

The investigators will prospectively study a total of 40 adult patients (> 18 years) divided into two subgroups: 20 laparoscopic surgery patients and 20 open surgery patients. After induction of anesthesia and neuromuscular blockade, all patients will be submitted to a recruitment maneuver in pressure-controlled ventilation (PCV) mode (PEEP = 20cmH2O, driving pressure = 20cmH2O, respiratory rate (RR) of 15 ipm and I:E ratio of 1:1) for 2 minutes followed by a decremental PEEP titration. The first step of the titration will start at a PEEP of 20 cmH2O and every 40 seconds PEEP will be decreased by 2 cmH2O, until a final PEEP of 4 cmH2O. A sub-sample of patients will have each step of the PEEP titration procedure recorded with an ultrasound and later evaluated by two different investigators. Optimal PEEP will be defined as that with the best compromise of atelectasis and overdistension as measured by EIT.

Patients in each subgroup will be randomized to one of two ventilatory strategies: (1) PEEP chosen by the PEEP titration procedure; (2) PEEP set at 4 cmH2O. After a new recruitment maneuver PEEP will be set at the designated value and the patient will be ventilated with an inspired oxygen fraction of 50% or greater in order to maintain peripheral oxygen saturation (SpO2) > 96%, a tidal volume of 6 mL/Kg and a respiratory rate to maintain an end tidal carbon dioxide (ETCO2) between 35-45.

All patients will have their global and regional pulmonary mechanics monitored by EIT throughout the anesthetic procedure to assess the degree of pulmonary atelectasis. After extubation, patients will be referred to the Radiology Department for a chest CT.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to general anesthesia for surgical procedure

Exclusion Criteria:

* Age < 18 years
* Thoracic surgery (any)
* ASA grade III or IV
* History of moderate/severe chronic obstructive pulmonary disease (COPD) or moderate/severe Asthma
* Moderate/severe restrictive lung disease
* Use of heart pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Optimal PEEP value | 6 minutes
  The PEEP value, for each patient, that produces the best possible compromise of lung collapse and lung hyperdistention during a PEEP titration procedure using EIT

SECONDARY OUTCOMES:
Pulmonary atelectasis | 2-5 hours
  The amount of atelectasis, in percentage of lung mass, evaluated by EIT during intraoperative period and by chest CT scan after extubation
Ultrasound evaluation | 6 minutes
  The use of ultrasound as a tool for PEEP titration intraoperatively compared to EIT

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim E Vieira, MD, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Tonelotto B, Pereira SM, Tucci MR, Vaz DF, Vieira JE, Malbouisson LM, Gay F, Simoes CM, Carvalho Carmona MJ, Monsel A, Amato MB, Rouby JJ, Costa Auler JO Jr. Intraoperative pulmonary hyperdistention estimated by transthoracic lung ultrasound: A pilot study. Anaesth Crit Care Pain Med. 2020 Dec;39(6):825-831. doi: 10.1016/j.accpm.2020.09.009. Epub 2020 Oct 17. PMID 33080407
- [Derived] Pereira SM, Tucci MR, Morais CCA, Simoes CM, Tonelotto BFF, Pompeo MS, Kay FU, Pelosi P, Vieira JE, Amato MBP. Individual Positive End-expiratory Pressure Settings Optimize Intraoperative Mechanical Ventilation and Reduce Postoperative Atelectasis. Anesthesiology. 2018 Dec;129(6):1070-1081. doi: 10.1097/ALN.0000000000002435. PMID 30260897